CLINICAL TRIAL: NCT04299022
Title: Safety, Efficacy, & Use of ViviGen Cellular Bone Matrix Allograft in Orthopaedic Fracture Care: A Multi-Center Prospective Registry and Retrospective Data Collection Study
Brief Title: Safety, Efficacy, & Use of ViviGen Cellular Bone Matrix Allograft in Orthopaedic Fracture Care
Status: Recruiting | Type: Observational
Sponsor: LifeNet Health (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-20-002
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Fractures, Bone; Nonunion of Fracture; Fractures, Open; Fractures, Ununited; Fracture, Tibial; Fracture of Femur; Fracture Arm
Keywords: fracture; nonunion; allograft
MeSH Terms: conditions — Fractures, Bone; Fractures, Ununited; Fractures, Open; Tibial Fractures; Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective Registry: Treatment for diagnoses of long bone non-union involving the tibia or femur and other nonunion diagnosis (i.e. clavicle, humerus, and femur) with Vivigen Cellular Bone Matrix
  Interventions: Other: Vivigen Cellular Bone Matrix
- Retrospective Data Collection: Treatment of diagnoses of long bone non-union involving the tibia or femur and other nonunion diagnosis (i.e. clavicle, humerus, and femur) with adjunct bone graft utilized in the acute, delayed, non-union and fusion settings.

INTERVENTIONS:
Other: Vivigen Cellular Bone Matrix — Allograft bone matrix
  Groups: Prospective Registry

SUMMARY:
Prospective registry and retrospective data collection study to assess the efficacy and safety of Vivigen Cellular Bone Matrix (Vivigen) in orthopaedic trauma patients who require bone grafting in the acute, delayed, non-union fracture as well as use in fusion procedure settings.

DETAILED DESCRIPTION:
The prospective registry study and retrospective data collection study is planned to assess the efficacy and safety of Vivigen Cellular Bone Matrix (Vivigen) in orthopaedic trauma patients who require bone grafting in the acute, delayed, non-union fracture as well as use in fusion procedure settings.

Patients will be assessed at hospital discharge, 6 weeks, 3 months, 6 months, 12 months and 24 months after treatment of a traumatic fracture with a bone graft.

ELIGIBILITY:
Prospective Cohort Inclusion Criteria:

* Any skeletally mature patient treated with Vivigen bone graft in the setting of an acute fracture, delayed, non-union or fusion setting will be eligible for inclusion.

Retrospective Cohort Inclusion Criteria:

- Any skeletally mature patient treated with adjunct bone graft in the setting of an acute fracture, delayed, non-union or fusion setting will eligible for inclusion.

Prospective Cohort Exclusion Criteria:

1. Patients unable to understand either an English or Spanish consent will be excluded.
2. Patients unable to consent secondary to dementia and/or other mental/psychiatric diagnoses will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospective data will be collected for up to 250 subjects across up to 7 academic medical centers that will receive Vivigen Cellular Bone Matrix for treatment of a fracture. Retrospective data will be collected for up to an additional 250 subjects that received a bone graft adjunct for treatment of a fracture.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Reintervention Rate | 24 months
  the proportion of patients requiring secondary intervention (return to the operating room) within twelve months after definitive wound closure

SECONDARY OUTCOMES:
Fusion Rate | 24 months
  Acute fracture, delayed union or nonunion rate as assessed with radiographs at 6 weeks, 3 months, 6 months, 12 months and 24 months
Patient Reported Outcome Measurement Information System (PROMIS) Scores | 24 months
  Patient reported outcome measures will be measured via PROMIS scoring tool (mental and physical). The PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For PROMIS measures, higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function). Thus a score of 60 is one standard deviation above the average referenced population.

CONTACTS AND LOCATIONS:
Overall Officials: Alyce Jones, Ph.D, Study Director — LifeNet Health
Locations (4):
- United States (4):
  - OrlandoHealth, Orlando, Florida
  - RWJBarnabas Health, Jersey City, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Sentara Hospitals, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No